CLINICAL TRIAL: NCT01980160
Title: Randomized Single-Blind Study of Nometex as an Adjunct to Standard Anti-emetics in Ovarian and Advanced Endometrial and Cervical Cancer Patients Who Receive Moderately to Highly Emetogenic Chemotherapy
Brief Title: Relief Band as an Adjunct to Antiemetic Therapy in Patients Who Receive Mod to Highly Emetogenic Chemotherapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not receive IRB approval from our institution therefore the study was closed.
Sponsor: Christiana Care Health Services (Other)
Collaborators: Neurowave Medical Technologies (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NMT-Nometex
Record Dates: First submitted 2013-10-14; First posted 2013-11-08 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Activated Nometex Device (Active Comparator): Nometex Device that is activated so will be sending electrical pulses to the median nerve which will travel through afferent nerve fibers to the emetic centers of the brain. It is in these areas that the neurotransmitters modulate signals going to the stomach via the Vagus nerve. These electrical signals normalize the stomach rhythms, thereby alleviating nausea and vomiting.
  Interventions: Device: Activated Nometex Device
- Unactivated Nometex Device (Sham Comparator): The Nometex device will not be activated and therefore have no effect on the nausea/vomiting associated with chemotherapy.
  Interventions: Device: Unactivated Nometex Device

INTERVENTIONS:
Device: Activated Nometex Device — Nometex Device that is activated so will be sending electrical pulses to the median nerve which will travel through afferent nerve fibers to the emetic centers of the brain. It is in these areas that the neurotransmitters modulate signals going to the stomach via the Vagus nerve. These electrical signals normalize the stomach rhythms, thereby alleviating nausea and vomiting.
  Arms: Activated Nometex Device
Device: Unactivated Nometex Device
  Other Names: Patients using this device will be given an unactivated Nometex device. It should be the same in appearance as the activated device.
  Arms: Unactivated Nometex Device

SUMMARY:
The primary study hypotheses are that, without increasing doses of breakthrough medications or device intolerance, the Nometex™ device worn for 5-days beginning with the day of chemotherapy administration in women with ovarian or advanced endometrial or cervical cancer will, as an adjunct to standard-of-care anti-emetics, reduce vomiting episodes, and reduce the severity of nausea.

The secondary hypotheses are that the Nometex™ device reduces acute (Day 1) emetic episodes, day 1 and days 2-5 severity of nausea, and delayed (days 2-5) emetic episodes without increasing doses of breakthrough medications or device intolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Women with ovarian (including fallopian tube) or advanced endometrial or cervical cancer
2. Chemotherapy-naïve or who have had previous chemotherapy exposure, but who have not yet received the first infusion
3. 18 years of age or older, and can provide cognizant informed consent presenting to the Helen F. Graham Cancer Center
4. ECOG Status of 0-2
5. Standardized Antiemetic Regimen

Exclusion Criteria:

1. Pre-existing or at-risk for a peripheral neuropathy in region of device placement
2. Implanted cardiac pace maker
3. Nickel or other metal allergies
4. Previous experience with median nerve/P6 stimulation
5. Receiving concurrent radiation therapy
6. Previous participants of this study will be excluded from future participation in this study.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2015-11 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Number of episodes of Vomiting | 1 month
  The primary outcome measure we are looking for is the number of vomiting episodes in patients with active wrist bands verse the sham wrist bands.
Severity of Nausea | 1 month
  One of the primary outcomes we are investigating is the severity of nausea in patients with active wrist bands verse the sham wrist bands.

SECONDARY OUTCOMES:
Acute Emetic Episodes | 1 day
  More specifically, the number of episodes of vomiting on Day 1.
Severity of nausea | 1 day
  The severity of acute nausea on day 1 of treatment.
Delayed severe nausea | 5 days
  The delayed number severe nausea episodes on days 2-5.
Delayed emetic episodes | 5 days
  Looking at the number of delayed emetic episodes during days 2-5 of treatment.
Rescue Medication Use | 1 month
  Will look at the use of rescue medication throughout treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Helen F. Graham Cancer Center, Newark, Delaware, United States

REFERENCES:
- [Background] Griffin AM, Butow PN, Coates AS, Childs AM, Ellis PM, Dunn SM, Tattersall MH. On the receiving end. V: Patient perceptions of the side effects of cancer chemotherapy in 1993. Ann Oncol. 1996 Feb;7(2):189-95. doi: 10.1093/oxfordjournals.annonc.a010548. PMID 8777177
- [Background] Osoba D, Zee B, Warr D, Latreille J, Kaizer L, Pater J. Effect of postchemotherapy nausea and vomiting on health-related quality of life. The Quality of Life and Symptom Control Committees of the National Cancer Institute of Canada Clinical Trials Group. Support Care Cancer. 1997 Jul;5(4):307-13. doi: 10.1007/s005200050078. PMID 9257427
- [Background] Lindley CM, Hirsch JD, O'Neill CV, Transau MC, Gilbert CS, Osterhaus JT. Quality of life consequences of chemotherapy-induced emesis. Qual Life Res. 1992 Oct;1(5):331-40. doi: 10.1007/BF00434947. PMID 1299465
- [Background] Laszlo J. Nausea and vomiting as major complications of cancer chemotherapy. Drugs. 1983 Feb;25 Suppl 1:1-7. doi: 10.2165/00003495-198300251-00002. PMID 6840017
- [Background] Campos D, Pereira JR, Reinhardt RR, Carracedo C, Poli S, Vogel C, Martinez-Cedillo J, Erazo A, Wittreich J, Eriksson LO, Carides AD, Gertz BJ. Prevention of cisplatin-induced emesis by the oral neurokinin-1 antagonist, MK-869, in combination with granisetron and dexamethasone or with dexamethasone alone. J Clin Oncol. 2001 Mar 15;19(6):1759-67. doi: 10.1200/JCO.2001.19.6.1759. PMID 11251007
- [Background] Birch R, Weaver CH, Carson K, Buckner CD. A randomized trial of once vs twice daily administration of intravenous granisetron with dexamethosone in patients receiving high-dose cyclophosphamide, thiotepa and carboplatin. Bone Marrow Transplant. 1998 Oct;22(7):685-8. doi: 10.1038/sj.bmt.1701412. PMID 9818697
- [Background] Navari RM, Reinhardt RR, Gralla RJ, Kris MG, Hesketh PJ, Khojasteh A, Kindler H, Grote TH, Pendergrass K, Grunberg SM, Carides AD, Gertz BJ. Reduction of cisplatin-induced emesis by a selective neurokinin-1-receptor antagonist. L-754,030 Antiemetic Trials Group. N Engl J Med. 1999 Jan 21;340(3):190-5. doi: 10.1056/NEJM199901213400304. PMID 9917226
- [Background] Shen J, Wenger N, Glaspy J, Hays RD, Albert PS, Choi C, Shekelle PG. Electroacupuncture for control of myeloablative chemotherapy-induced emesis: A randomized controlled trial. JAMA. 2000 Dec 6;284(21):2755-61. doi: 10.1001/jama.284.21.2755. PMID 11105182
- [Background] Treish I, Shord S, Valgus J, Harvey D, Nagy J, Stegal J, Lindley C. Randomized double-blind study of the Reliefband as an adjunct to standard antiemetics in patients receiving moderately-high to highly emetogenic chemotherapy. Support Care Cancer. 2003 Aug;11(8):516-21. doi: 10.1007/s00520-003-0467-3. Epub 2003 Jun 27. PMID 12836088
- [Background] Gralla RJ, Osoba D, Kris MG, Kirkbride P, Hesketh PJ, Chinnery LW, Clark-Snow R, Gill DP, Groshen S, Grunberg S, Koeller JM, Morrow GR, Perez EA, Silber JH, Pfister DG. Recommendations for the use of antiemetics: evidence-based, clinical practice guidelines. American Society of Clinical Oncology. J Clin Oncol. 1999 Sep;17(9):2971-94. doi: 10.1200/JCO.1999.17.9.2971. No abstract available. PMID 10561376
- [Background] Oyama H, Kaneda M, Katsumata N, Akechi T, Ohsuga M. Using the bedside wellness system during chemotherapy decreases fatigue and emesis in cancer patients. J Med Syst. 2000 Jun;24(3):173-82. doi: 10.1023/a:1005591626518. PMID 10984871
- [Background] Wickham R. Evolving treatment paradigms for chemotherapy-induced nausea and vomiting. Cancer Control. 2012 Apr;19(2 Suppl):3-9. doi: 10.1177/107327481201902s02. PMID 22488022
- [Background] Schwartzberg LS. Chemotherapy-induced nausea and vomiting: which antiemetic for which therapy? Oncology (Williston Park). 2007 Jul;21(8):946-53; discussion 954, 959, 962 passim. PMID 17715696
- [Background] Sigsgaard T, Herrstedt J, Handberg J, Kjaer M, Dombernowsky P. Ondansetron plus metopimazine compared with ondansetron plus metopimazine plus prednisolone as antiemetic prophylaxis in patients receiving multiple cycles of moderately emetogenic chemotherapy. J Clin Oncol. 2001 Apr 1;19(7):2091-7. doi: 10.1200/JCO.2001.19.7.2091. PMID 11283143
- [Background] Herrington JD, Kwan P, Young RR, Lagow E, Lagrone L, Riggs MW. Randomized, multicenter comparison of oral granisetron and oral ondansetron for emetogenic chemotherapy. Pharmacotherapy. 2000 Nov;20(11):1318-23. doi: 10.1592/phco.20.17.1318.34894. PMID 11079280
- [Background] Osowski CL, Dix SP, Lynn M, Davidson T, Cohen L, Miyahara T, Sexauer MC, Joyce R, Yeager A, Wingard JR. An open-label dose comparison study of ondansetron for the prevention of emesis associated with chemotherapy prior to bone marrow transplantation. Support Care Cancer. 1998 Nov;6(6):511-7. doi: 10.1007/s005200050206. PMID 9833299